CLINICAL TRIAL: NCT04540146
Title: Evaluation of T Helper Cytokines in Intraabdominal Ascites in End Stage Colorectal Cancers
Brief Title: T Helper Cytokines in End Stage Colorectal Cancers
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD, Istanbul Training and Research Hospital
Other Study IDs: Colorectal cytokine
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer
Keywords: Ascites; T cell; Flow-cytometry; Cytokine
MeSH Terms: conditions — Colorectal Neoplasms; Ascites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: End Stage Colorectal Cancer patients with intraabdominal ascites
  Interventions: Diagnostic Test: Flow-Cytometric analysis
- Control: Congestive heart failure and liver cirrhosis patient who had intraabdominal ascites
  Interventions: Diagnostic Test: Flow-Cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow-Cytometric analysis — IL-2, 4, 5, 6, 9, 10, 13, 17A, 17F, 22, IFN-γ and TNF-α levels in the intraabdominal ascites

SUMMARY:
Colorectal cancers are the third most common type of cancer in the world. Peritoneal carcinomatosis and intraabdominal acid development occur in advanced stages of colorectal cancers.

It is known that the immune system plays an important role in tumor development or tumor eradication. Differentiation of T cells towards Th2 and regulatory T cells is also reported to be effective in tumor progression.

Among the mechanisms of escape from the immune system, changes in the tumor microenvironment play an important role. The role of regulatory T lymphocytes, a subgroup of T cells that play a regulatory role by suppressing the function of other T lymphocytes, is to reduce the chronic immune response against viruses, tumors and patients's own antigens. The common feature of all Tregs is that they secrete one or more anti-inflammatory molecules such as IL-10, TGFβ or IL-35. High levels of Tregs have been found in peripheral blood, tumor tissue and lymph nodes in patients with malignancy.

In our study, it is aimed to evaluate whether there is a difference in intraabdominal ascites fluid T helper cytokine levels in patients with end-stage colorectal cancers compared to patients without malignancy.

DETAILED DESCRIPTION:
Colorectal cancers are the third most common type of cancer in the world. Peritoneal carcinomatosis and intraabdominal ascites development occur in advanced stages of colorectal cancers.

It is known that the immune system plays an important role in tumor development or tumor eradication. Differentiation of T cells towards Th2 and regulatory T cells is also reported to be effective in tumor progression.

Among the mechanisms of escape from the immune system, changes in the tumor microenvironment play an important role. The role of regulatory T lymphocytes, a subgroup of T cells that play a regulatory role by suppressing the function of other T lymphocytes, is to reduce the chronic immune response against viruses, tumors and patient's own antigens. The common feature of all Tregs is that they secrete one or more anti-inflammatory molecules such as IL-10, TGFβ or IL-35. High levels of Tregs have been found in peripheral blood, tumor tissue and lymph nodes in patients with malignancy.

The role of the immune system in colorectal cancers has been demonstrated with the effects of tumor-infiltrating lymphocytes (TIL) and immune control points on TILs or immune control point ligands on patient survival, especially in recent studies. Studies in the literature usually include immunological examinations of patient blood or tumor tissue.

There are many publications in the literature evaluating immunological markers from ascites fluid samples for various reasons. In these studies, T and B cell subtypes were examined from ascites fluid samples taken from patients with ascites, especially ovarian cancer and liver cirrhosis. In the only study on gastrointestinal cancers, immunophenotyping was performed in intraabdominal ascites and blood in 22 advanced gastrointestinal tumor patients and some cell subgroups were associated with worse clinical outcome. In the literature, there is no study on cytokine analysis from intra-abdominal ascites fluids specific to colorectal cancer.

In our study, it is aimed to evaluate whether there is a difference in intraabdominal ascites fluid cytokine level in patients with end-stage colorectal patients compared to patients without malignancy.

ELIGIBILITY:
Inclusion Criteria:

* End stage Colorectal Cancer patients

Exclusion Criteria:

* Another synchronous tumor with colorectal cancer
* HIV patients
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The end stage colorectal cancer patients with intraabdominal ascites will be the case group.
  Also congestive heart failure and liver cirrhosis patients with intraabdominal ascites will be the control group
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
cytokine levels | 3 months
  IL-2, 4, 5, 6, 9, 10, 13, 17A, 17F, 22, IFN-γ and TNF-α levels

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Ufuk Oguz Idiz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Syed Khaja AS, Toor SM, El Salhat H, Ali BR, Elkord E. Intratumoral FoxP3+Helios+ Regulatory T Cells Upregulating Immunosuppressive Molecules Are Expanded in Human Colorectal Cancer. Front Immunol. 2017 May 26;8:619. doi: 10.3389/fimmu.2017.00619. eCollection 2017. PMID 28603527
- [Background] Yoshida N, Kinugasa T, Miyoshi H, Sato K, Yuge K, Ohchi T, Fujino S, Shiraiwa S, Katagiri M, Akagi Y, Ohshima K. A High RORgammaT/CD3 Ratio is a Strong Prognostic Factor for Postoperative Survival in Advanced Colorectal Cancer: Analysis of Helper T Cell Lymphocytes (Th1, Th2, Th17 and Regulatory T Cells). Ann Surg Oncol. 2016 Mar;23(3):919-27. doi: 10.1245/s10434-015-4923-3. Epub 2015 Nov 12. PMID 26564244
- [Background] Nakano M, Ito M, Tanaka R, Yamaguchi K, Ariyama H, Mitsugi K, Yoshihiro T, Ohmura H, Tsuruta N, Hanamura F, Sagara K, Okumura Y, Nio K, Tsuchihashi K, Arita S, Kusaba H, Akashi K, Baba E. PD-1+ TIM-3+ T cells in malignant ascites predict prognosis of gastrointestinal cancer. Cancer Sci. 2018 Sep;109(9):2986-2992. doi: 10.1111/cas.13723. PMID 30187676